CLINICAL TRIAL: NCT03450707
Title: Thiamine as a Metabolic Resuscitator After Cardiac Arrest
Acronym: THACA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMB recommendation based on differing mortality in a subgroup analysis
Sponsor: Michael Donnino (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Michael Donnino, Associate Professor of Medicine and Emergency Medicine, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017P000245; 1R01HL136705-01 (NIH)
Record Dates: First submitted 2018-02-21; First posted 2018-03-01 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; post-arrest
MeSH Terms: conditions — Heart Arrest | interventions — Thiamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomization list was prepared by an independent statistician using 1:1 randomization in blocks of four. This list will be provided to the research pharmacy, and the research pharmacy will be the only unblinded people involved with the study, and will have no patient contact or role in the analysis or other aspects of the study. Thiamine is colorless and odorless, and the 500mg dose is mixed in 100mL of normal saline. Placebo will be 100mL of normal saline and is indistinguishable in appearance from thiamine. Study team, clinical team and patient and family will all be blind to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Thiamine (Experimental): Patients randomized to the thiamine arm will receive thiamine 500mg in 100mL of normal saline intravenously every 12 hours for 5 doses. Patients will be connected to a noninvasive monitor for measurement of global oxygen consumption (VO2) for at least 48 hours or until extubated, whichever comes first. Blood will be drawn at 0,6,12,24,72 and 168 hours for measurement of lactate, thiamine level, pyruvate dehydrogenase, NSE, S100 and other markers of organ injury. CPC-E score will be assessed prior to hospital discharge and at 30 and 90 days to evaluate differences in neurologic and functional impairment.
  Interventions: Drug: Thiamine 500 mg IV
- Placebo (Placebo Comparator): Patients randomized to placebo will receive 100mL normal saline intravenously every 12 hours for 5 doses. All other aspects of the protocol will be the same as in the experimental arm. Patients will be connected to a noninvasive monitor for measurement of global oxygen consumption (VO2) for at least 48 hours or until extubated, whichever comes first. Blood will be drawn at 0,6,12,24,72 and 168 hours for measurement of lactate, thiamine level, pyruvate dehydrogenase, NSE, S100 and other markers of organ injury. CPC-E score will be assessed prior to hospital discharge and at 30 and 90 days to evaluate differences in neurologic and functional impairment.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Thiamine 500 mg IV — Thiamine hydrochloride (vitamin B1) 500mg IV will be given every 12 hours for 5 doses in the experimental arm.
  Other Names: vitamin B1
  Arms: Thiamine
Other: Placebo — 100mL of intravenous normal saline will be given every 12hours for 5 doses in the placebo arm
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo controlled study to investigate the effect of intravenous thiamine (vitamin B1) on lactate, cellular oxygen consumption, global oxygen consumption and biomarkers of neurologic injury after out-of-hospital cardiac arrest (OHCA). .

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled study to investigate the effect of intravenous thiamine (vitamin B1) on lactate, cellular oxygen consumption, global oxygen consumption and biomarkers of neurologic injury after out-of-hospital cardiac arrest (OHCA). Patients who have sustained return of spontaneous circulation (ROSC) after OHCA and have a lactate of 3 or greater will be eligible for the study. Enrolled patients will be randomized to intravenous thiamine 500mg twice daily for 5 doses or matching placebo (100cc normal saline). Blood will be drawn at several time points and patients will be connected to a noninvasive monitor for continuous measurement of global oxygen consumption. The primary endpoint is change in lactate level. Secondary endpoints include change in pyruvate dehydrogenase activity, change in cellular and global oxygen consumption, change in NSE and S100 (biomarkers of neurologic injury) and CPC-E score (a score that assesses neurologic and functional impairment) at hospital discharge, 30 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age ≥ 18 years)
* Cardiac arrest occurring with sustained (> 20 minutes) return of spontaneous circulation (ROSC)
* Within 4.5 hours of cardiac arrest event
* Lactate >/=3

Exclusion Criteria:

* Clinical indication for thiamine administration (alcoholism, known or highly suspected deficiency) or treatment with thiamine beyond the amount found in a standard multivitamin within the last 10 days
* Traumatic etiology of arrest
* Comfort measures only or anticipated withdrawal of support within 24 hours
* Protected populations (pregnant women, prisoners)
* Known allergy to thiamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-05-06 (Actual); Primary Completion 2022-02-19 (Actual); Study Completion 2022-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thiamine | Placebo
Started (93 is the total number of patients who were randomized to either thiamine or placebo:47 randomized to thiamine, 46 randomized to placebo. But 7/47 randomized to thiamine did not receive the intervention, and 10/46 randomized to placebo did not receive the placebo, resulting in final numbers of 40 patients who received thiamine and 36 patients who received placebo. A granular breakdown of the reasons for not having received the intervention is given in the "reason not completed" field.) | 47 | 46
Completed | 40 | 36
Not Completed | 7 | 10
Not completed — Outside enrollment window | 4 | 1
Not completed — Death | 1 | 0
Not completed — Indication for thiamine | 1 | 1
Not completed — Evidence of traumatic brain injury | 1 | 0
Not completed — Following commands | 0 | 3
Not completed — Lactate < 3.5 | 0 | 2
Not completed — Rearrest with ECMO | 0 | 1
Not completed — Indication for thiamine + head CT results | 0 | 1
Not completed — Family/patient goals of care | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thiamine | Placebo | Total
Number analyzed (Participants) | 40 | 36 | 76
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68.5 [58.0 to 79.5] | 65.5 [58.0 to 79.0] | 66.5 [58.0 to 79.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 25 | 20 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 14 | 20 | 34
  Unknown or Not Reported | 24 | 14 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 10 | 17 | 27
  Race: Black | 6 | 3 | 9
  Race: Asian | 3 | 0 | 3
  Race: Other | 0 | 2 | 2
  Race: Unknown | 21 | 14 | 35
Initial Rhythm [Count of Participants; unit: Participants]
  Pulseless electrical activity | 15 | 13 | 28
  Asystole | 9 | 10 | 19
  Ventricular Fibrillation | 6 | 5 | 11
  Pulseless Ventricular Tachycardia | 3 | 1 | 4
  Unknown Shockable | 4 | 5 | 9
  Unknown Non-Shockable | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Lactate
Description: Blood Lactate Over Time
Time Frame: 24 hours
Population: Seventeen patients (six in the placebo arm and eleven in the thiamine arm) missing 24-hour lactate as they had expired by this timepoint.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 29 | 30
mmol/L | 1.8 [1.2 to 2.4] | 2.2 [1.4 to 2.5]
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other; p = 0.72, Mixed Models Analysis — Mixed model controlling for repeated measures within patients used to get a mean difference in lactate between the thiamine and placebo groups at 24 hours. Lactate imputed using a penalty (20pc increase) for patients who expired; P-value is for the comparison at 24 hours from the mixed model (i.e, not a global p-value); Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-1.82 to 2.50]

2. Secondary Outcome: Global Oxygen Consumption
Description: Global Oxygen Consumption over Time
Time Frame: 48 hours
Population: Only 12 patients in the thiamine group and 18 patients in the placebo group had atleast 60 minutes of metabolic data in the first 48 hours after study drug administration
Measure: Mean (Standard Deviation); unit: Area under the Curve VO2 (mL/kg/min)
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 12 | 18
Area under the Curve VO2 (mL/kg/min) | 3.52 (1.50) | 3.93 (1.05)
Statistical Analysis 1: Comparison: Thiamine vs Placebo; As AUC-VO2s turned out to be normally distributed, we used a linear regression model to compare mean AUC-VO2s between treatment groups controlling for average temperature; Test type: Other; p = 0.43, Regression, Linear; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-1.34 to 0.58]

3. Secondary Outcome: Lactate
Description: Absolute Blood Level of Lactate
Time Frame: 72 hours
Population: Thirty-two patients (thirteen in the placebo arm and nineteen in the thiamine arm) missing 72-hour lactate as they had expired prior to the 72-hour timepoint.
  In addition, two more patients in the placebo arm alive at 72 hours were missing 72-hour lactate due to health care provider request/patient refusal.
  No imputation was done for this secondary outcome.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 21 | 21
mmol/L | 1.3 [0.9 to 1.6] | 1.3 [0.9 to 1.5]
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Wilcoxon rank-sum test, testing the null hypothesis that there is no difference in the distribution of 72-hour lactates between thiamine and placebo groups; Test type: Other; p = 0.88, Wilcoxon (Mann-Whitney); No parameter estimated other than p-value = 0.88 from Wilcoxon rank-sum test

4. Secondary Outcome: Pyruvate Dehydrogenase (PDH) Specific Activity
Description: Absolute PDH specific activity value
Time Frame: 72 hours
Population: Only 20 patients from the thiamine group and 15 patients from the placebo group were alive and had PDH specific activity available at 72 hours.
Measure: Median (Inter-Quartile Range); unit: Ratio [PDH activity/ln(PDH quantity)]
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 20 | 15
Ratio [PDH activity/ln(PDH quantity)] | 1.55 [0.88 to 2.11] | 0.97 [0.78 to 1.60]
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other; p = 0.072, Mixed Models Analysis — Mixed model controlling for repeated measures within patients used to get a mean difference in PDH specific activity between the thiamine and placebo groups at 72 hours; P-value is the global p-value from the mixed model. P-value is obtained from a model that uses a log-transformed version of the variable; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [0.01 to 0.80]

5. Secondary Outcome: Pyruvate Dehydrogenase (PDH) Activity
Description: Absolute PDH Activity Value
Time Frame: 72 hours
Population: Only 20 patients from the thiamine group and 16 patients from the placebo group were alive and had PDH activity available at 72 hours.
Measure: Median (Inter-Quartile Range); unit: mini OD unit/min/mg protein
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 20 | 16
mini OD unit/min/mg protein | 8.63 [4.93 to 12.90] | 5.65 [4.77 to 9.38]
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other; p = 0.044, Mixed Models Analysis — Mixed model controlling for repeated measures within patients used to get a mean difference in PDH activity between the thiamine and placebo groups at 72 hours; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [0.1 to 4.7]

6. Secondary Outcome: Pyruvate Dehydrogenase (PDH) Quantity
Description: Absolute PDH Quantity. Please note that the measurement of Absolute PDH Quantity is done using a relative quantity assay, and that PDH is an enzyme and not a stable protein; therefore the units of measure cannot be provided in "mg" and are instead listed in "mini OD unit/min/mg protein".
Time Frame: 72 hours
Population: Only 20 patients from the thiamine group and 15 patients from the placebo group were alive and had PDH quantity available at 72 hours.
Measure: Median (Inter-Quartile Range); unit: mini OD unit/min/mg protein
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 20 | 15
mini OD unit/min/mg protein | 588.05 [291.31 to 1080.94] | 695.55 [437.94 to 999.09]
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other; p = 0.828, Mixed Models Analysis — Mixed model controlling for repeated measures within patients used to get a mean difference in PDH quantity between the thiamine and placebo groups at 72 hours; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -48.5, 95% CI 2-sided [-297.0 to 200.0]

7. Secondary Outcome: Mortality
Description: Mortality in the study assessed at three timepoints.
Time Frame: will be assessed at hospital discharge and up to 30 and 90 days.
Population: For 90-day mortality, two patients from the placebo arm were not reachable for follow-up and thus are missing this information.
Measure: Count of Participants; unit: Participants
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 40 | 36
Participants
  Discharge mortality | 30 | 23
  30-day mortality | 30 | 24
  90-day mortality: number analyzed (Participants) | 40 | 34
  90-day mortality | 30 | 24

8. Secondary Outcome: Favorable Cerebral Performance Category (CPC)
Description: Count/Proportion of Patients Scoring a Favorable CPC, defined as a score of 1 or 2.
  Cerebral performance category scores range from 1-5. Lower scores mean better outcomes.
Time Frame: will be assessed up to 30 and 90 days
Population: Two patients, both from placebo arm, did not have 30 day CPC scores available. Four patients, all from the placebo arm, did not have 90 day CPC scores available.
Measure: Count of Participants; unit: Participants
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 40 | 36
Participants
  Favorable Discharge CPC (1-2) | 8 | 10
  Favorable 30-day CPC (1-2): number analyzed (Participants) | 40 | 34
  Favorable 30-day CPC (1-2) | 9 | 9
  Favorable 90-day CPC (1-2): number analyzed (Participants) | 40 | 32
  Favorable 90-day CPC (1-2) | 9 | 7

9. Secondary Outcome: Sequential Organ Failure Assessment (SOFA) Score
Description: SOFA score over time.
  SOFA score: Sequential Organ Failure Assessment Score, ranges from 0-24, higher scores mean worse outcomes.
Time Frame: over 72 hours
Population: 13 patients in the placebo arm and 19 patients in the thiamine arm missing 72-hour SOFA scores as they had expired by this timepoint.
  3 additional patients in the placebo arm were alive at 72-hours but are still missing 72-hour SOFA scores because one or more component scores required to calculate the SOFA scores were missing.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 21 | 20
score on a scale | 9 [7 to 12] | 6 [4 to 9]
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other; p = 0.10, Mixed Models Analysis — Mixed model controlling for repeated measures within patients used to get a mean difference in SOFA scores between the thiamine and placebo groups at 72 hours; P-value is the global p-value from the mixed model; Mean Difference (Final Values) = 2.34, 95% CI 2-sided [0.47 to 4.22]

10. Secondary Outcome: Acute Renal Failure
Description: Determined using the Kidney Disease Improving Global Outcomes (KDIGO) criteria for Stage 3 acute kidney injury/kidney failure.
Time Frame: First 7 days following Arrest
Population: Three patients from the placebo arm and one from the thiamine arm were excluded from the renal failure analyses due to pre-arrest end-stage renal disease requiring dialyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 39 | 33
Participants | 9 | 3

11. Secondary Outcome: Cellular Oxygen Consumption
Description: Absolute Cellular Oxygen Consumption Rate: We use two measures to capture Oxygen Consumption Rate; the basal respiration and the maximal respiration.
Time Frame: 0 hours and 24 hours.
Population: Two patients from the thiamine group had a thiamine value >1200 and were excluded.
Measure: Median (Inter-Quartile Range); unit: pmol/min/mg protein
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 38 | 36
pmol/min/mg protein
  Basal respiration-0 hours | 5.6 [4.3 to 7.8] | 4.8 [3.2 to 7.9]
  Maximal respiration-0 hours | 19.3 [7.9 to 36.1] | 11.9 [6.8 to 30.3]
  Basal respiration-24 hours | 5.5 [2.6 to 6.3] | 4.7 [3.4 to 9.3]
  Maximal respiration-24 hours | 14.7 [10.4 to 25.1] | 16.1 [11.5 to 34.3]
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other; p = 0.43, Mixed Models Analysis — Mixed model controlling for repeated measures within patients used to get a mean difference in Basal Respiration between the thiamine and placebo groups at 24 hours; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-3.6 to 1.6] — Mean difference uses a non-logged version of the variable

12. Secondary Outcome: Creatinine
Description: Creatinine over Time
Time Frame: 72 hours
Population: Thirty-two patients (thirteen in the placebo arm and nineteen in the thiamine arm) missing 72-hour creatinine as they had expired prior to the 72-hour timepoint.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 21 | 23
mg/dL | 1.9 [0.9 to 2.8] | 1.1 [0.8 to 1.9]
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other; p = 0.02, Mixed Models Analysis — Mixed model controlling for repeated measures within patients used to get a mean difference in creatinine between the thiamine and placebo groups at 72 hours; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [-0.27 to 1.78]

13. Secondary Outcome: Biomarkers of Neurologic Injury
Description: S100 and NSE levels at various time points
Time Frame: various time points over 7 days
Population: Biomarker assays not run in the laboratory at this time
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored upto 90 days; Serious and/or Other (Not Including Serious) Adverse Events assessed from enrollment to time of discharge, an average of one week.
Arm/Group | Thiamine | Placebo
All-Cause Mortality (participants affected / at risk) | 30/40 | 24/36
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/36
Other Adverse Events (participants affected / at risk) | 0/40 | 0/36

LIMITATIONS AND CAVEATS:
The study was stopped early by the Data Safety and Monitoring Board (DSMB) due to a signal of increased mortality in the thiamine group with a lactate > 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT03450707/Prot_SAP_001.pdf